CLINICAL TRIAL: NCT06541301
Title: PICC-ports Versus Chest - Ports for Long Term Chemotherapy Deliverance in Oncology Patients Affected by Solid Tumors. A Prospective, Randomized Multicentric, Non Inferiority, Phase III Trial.
Brief Title: PICC-ports Versus Chest - Ports for Long Term Chemotherapy Deliverance in Oncology Patients
Acronym: PICCHEST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: L2-113
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-07

CONDITIONS: Solid Tumor
Keywords: Solid Tumor; Chest-ports; Peripherally Inserted Central Catheters-ports

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, multicenter, open-label, non-inferiority clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PICC-port arm (Experimental): Implantation of a PICC-port device
  Interventions: Device: PICC-port
- Chest-port arm (Active Comparator): Implantation of a Chest-port device
  Interventions: Device: Chest-port

INTERVENTIONS:
Device: PICC-port — Implantation of a PICC-port device by a dedicated PICC team member following predefined evidence-based international guidelines and protocols
  Arms: PICC-port arm
Device: Chest-port — Implantation of a Chest-port device by expert physicians or certified expert nurses, following predefined evidence-based international guidelines and protocols
  Arms: Chest-port arm

SUMMARY:
Central venous access devices are extensively used in oncology patients. The current standard is represented by devices inserted by direct ultrasound guided cannulation of deep veins of supra/infraclavicular area with a reservoir placed in a subcutaneous pocket of the upper chest wall ("chest-ports"). More recently, PICC (Peripherally Inserted Central Catheters)-ports have been proposed as an alternative to chest-ports.

Aim of this study is to demonstrate the non-inferiority of PICC ports compared to thoracic ports in terms of efficacy and safety.

DETAILED DESCRIPTION:
Central venous access devices are extensively used in oncology patients who need safe deliverance of chemotherapeutic agents and drugs, transfusion of blood and blood products, and performance of laboratory tests, in solid as well as hematologic malignancies. These devices are mostly inserted by direct ultrasound guided cannulation of deep veins of supra/infraclavicular area and the reservoir is placed in a subcutaneous pocket of the upper chest wall ("chest-ports"). More recently, PICC (Peripherally Inserted Central Catheters)-ports have been proposed as a safe and effective alternative to chest-ports, claiming lower invasiveness, easier insertion and better patients' compliance. In PICC-ports a small reservoir is placed in a subcutaneous pocket located in the mid-third of the upper arm.

Since these feelings are currently based only on limited retrospective studies, aim of this randomized multicenter trial is to demonstrate the non-inferiority of PICC ports (experimental arm) compared to thoracic ports (control arm, as the current reference standard) in terms of efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 Age ≤ 75 yrs
* Histologic diagnosis of a solid tumour
* Need for intravenous , long term (> 3 months), intermittent chemotherapy (either adjuvant or palliative)
* Eastern Cooperative Oncology Group (ECOG) Performance Status: 0-2

Exclusion Criteria:

* Active infections
* Coagulopathy, defined as platelet count < 50,000/μL and/or Prothrombin time (PT)/International Normalized Ratio (INR) > 1.5
* Chronic severe renal failure, stage 3b-4-5 or imminent need for a dialysis fistula
* Any conditions contraindicating chemotherapy treatments, as valued by treating oncologist
* Life expectancy < 6 months, as valued by treating oncologist
* Inability to give an informed consent and/or history of psychiatric or addictive disorder or other medical condition that, in the opinion of the investigator, would preclude the patient from meeting the trial requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 852 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of device failures | 6 months
  Number of unscheduled removal of the device due to complications

SECONDARY OUTCOMES:
Incidence of adverse events associated to device | 6 months
  Number of adverse events associated with the implantation and use of the device that do not necessitate its removal

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Biffi, MD, Principal Investigator — European Istitute of Oncology
Locations (3):
- Italy (3):
  - CRO (Centro di Riferimento Oncologico), Aviano
  - Ospedale Careggi, Florence
  - European Institute of Oncology, Milan

REFERENCES:
- [Background] Gallieni M, Pittiruti M, Biffi R. Vascular access in oncology patients. CA Cancer J Clin. 2008 Nov-Dec;58(6):323-46. doi: 10.3322/CA.2008.0015. Epub 2008 Oct 29. PMID 18971486
- [Background] Biffi R, Pozzi S, Bonomo G, Della Vigna P, Monfardini L, Radice D, Rotmensz N, Zampino MG, Fazio N, Orsi F. Cost effectiveness of different central venous approaches for port placement and use in adult oncology patients: evidence from a randomized three-arm trial. Ann Surg Oncol. 2014 Nov;21(12):3725-31. doi: 10.1245/s10434-014-3784-5. Epub 2014 May 20. PMID 24841352
- [Background] Biffi R, Toro A, Pozzi S, Di Carlo I. Totally implantable vascular access devices 30 years after the first procedure. What has changed and what is still unsolved? Support Care Cancer. 2014 Jun;22(6):1705-14. doi: 10.1007/s00520-014-2208-1. PMID 24659216
- [Background] Bertoglio S, Cafiero F, Meszaros P, Varaldo E, Blondeaux E, Molinelli C, Minuto M. PICC-PORT totally implantable vascular access device in breast cancer patients undergoing chemotherapy. J Vasc Access. 2020 Jul;21(4):460-466. doi: 10.1177/1129729819884482. Epub 2019 Nov 1. PMID 31674857
- [Background] Bertoglio S, Annetta MG, Brescia F, Emoli A, Fabiani F, Fino M, Merlicco D, Musaro A, Orlandi M, Parisella L, Pinelli F, Reina S, Selmi V, Solari N, Tricarico F, Pittiruti M. A multicenter retrospective study on 4480 implanted PICC-ports: A GAVeCeLT project. J Vasc Access. 2022 Jan 17:11297298211067683. doi: 10.1177/11297298211067683. Online ahead of print. PMID 35034480
- [Background] Nickel B, Gorski L, Kleidon T, Kyes A, DeVries M, Keogh S, Meyer B, Sarver MJ, Crickman R, Ong J, Clare S, Hagle ME. Infusion Therapy Standards of Practice, 9th Edition. J Infus Nurs. 2024 Jan-Feb 01;47(1S Suppl 1):S1-S285. doi: 10.1097/NAN.0000000000000532. No abstract available. PMID 38211609
- [Background] Li G, Zhang Y, Ma H, Zheng J. Arm port vs chest port: a systematic review and meta-analysis. Cancer Manag Res. 2019 Jul 3;11:6099-6112. doi: 10.2147/CMAR.S205988. eCollection 2019. PMID 31308748
- [Background] Liu Y, Li LL, Xu L, Feng DD, Cao Y, Mao XY, Zheng J, Jin F, Chen B. Comparison between Arm Port and Chest Port for Optimal Vascular Access Port in Patients with Breast Cancer: A Systematic Review and Meta-Analysis. Biomed Res Int. 2020 Feb 13;2020:9082924. doi: 10.1155/2020/9082924. eCollection 2020. PMID 32104708
- [Background] Annetta MG, Bertoglio S, Biffi R, Brescia F, Giarretta I, Greca A, Panocchia N, Passaro G, Perna F, Pinelli F, Pittiruti M, Prisco D, Sanna T, Scoppettuolo G. Management of antithrombotic treatment and bleeding disorders in patients requiring venous access devices: A systematic review and a GAVeCeLT consensus statement. J Vasc Access. 2022 Jul;23(4):660-671. doi: 10.1177/11297298211072407. Epub 2022 May 9. PMID 35533088
- [Background] Biffi R, Orsi F, Pozzi S, Pace U, Bonomo G, Monfardini L, Della Vigna P, Rotmensz N, Radice D, Zampino MG, Fazio N, de Braud F, Andreoni B, Goldhirsch A. Best choice of central venous insertion site for the prevention of catheter-related complications in adult patients who need cancer therapy: a randomized trial. Ann Oncol. 2009 May;20(5):935-40. doi: 10.1093/annonc/mdn701. Epub 2009 Jan 29. PMID 19179550